CLINICAL TRIAL: NCT01829022
Title: Multi-center Prospective Study on Embryonic-Natural Orifice Transumbilical Endoscopic Surgery for Myomectomy With Traction of Multidirectional Sutures
Brief Title: Multi-center Prospective Study on E-NOTES for Myomectomy With Traction of Multidirectional Sutures
Acronym: E-NOTES
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: The Catholic University of Korea (Other); Saint Vincent's Hospital, Korea (Other); Incheon St.Mary's Hospital (Other); Kyung Hee University Hospital at Gangdong (Other); Keimyung University Dongsan Medical Center (Other); Korea University Guro Hospital (Other); Korea University Anam Hospital (Other); Cheil General Hospital and Women's Healthcare Center (Other); National Health Insurance Service Ilsan Hospital (Other); Seoul National University Bundang Hospital (Other); Seoul National University Hospital (Other); Samsung Medical Center (Other); Soonchunhyang University Hospital (Other); Ajou University (Other); Pusan National University Yangsan Hospital (Other); Severance Hospital (Other); Asan Medical Center (Other); Ewha Womans University Mokdong Hospital (Other); Inje University (Other); CHA University (Other); Kyungpook National University Hospital (Other); Hallym University Medical Center (Other); Hanyang University (Other)
Responsible Party: Principal Investigator, Myong Cheol Lim, Senior researcher, National Cancer Center, Korea
Other Study IDs: NCCNCS-13-MAR
Record Dates: First submitted 2013-03-27; First posted 2013-04-11 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Myoma
Keywords: Myoma; Uterine myomectomy
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- E-NOTES: Embryonic-Natural Orifice Transumbilical Endoscopic Surgery for Myomectomy with Traction of Multidirectional Sutures
  Interventions: Procedure: E-NOTES

INTERVENTIONS:
Procedure: E-NOTES — Embryonic-Natural Orifice Transumbilical Endoscopic Surgery for Myomectomy with Traction of Multidirectional Sutures
  Other Names: Embryonic-Natural Orifice Transumbilical Endoscopic Surgery

SUMMARY:
Primary objectives : To investigate technical feasibility and postoperative morbidity after E-NOTES for Myomectomy with Traction of Multidirectional Sutures

Secondary objectives : To investigate postoperative pain after E-NOTES for Myomectomy with Traction of Multidirectional Sutures by clinical variables such as incision size, type of port, size and number of myoma, or operation time.

DETAILED DESCRIPTION:
* Leiomyoma is a common benign tumor of the smooth muscle cells of the myometrium.1 It can cause several symptoms such as abnormal vaginal bleeding, pain, or urinary symptoms according to size and location. Steadily, lesser invasive surgeries have been preferred for such benign disease (laparotomy, laparoscopy, and then single-port surgery).2,3
* However, these minimal approaches, laparoscopic morcellation of preoperatively suspicious leimyoma, have the potential risk of peritoneal seeding of postoperative diagnosed leiomyosarcoma in the pathological examination.4 Currently, safe morcellation is also required during myomectomy while using a lesser invasive surgical approach such as single-port surgery or natural orifice transumbilical endoscopic surgery (NOTES).
* During single-port surgery or embryonic NOTES (E-NOTES) via an umbilicus, handling of myoma into different directions could be quite a big challenge. Fortunately, myoma is enough hard to pull with string and has a tendency not to rupture during manipulation of these strings.
* These concepts lead to traction of anchoring sutures during E-NOTES for myomectomy applied in the current case. Safe morcellation could be guaranteed, because direction morcellation via an umbilicus is possible in an endobag.
* This useful and safe surgical approach needs to be confirmed in multi-centers in terms of feasibility and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Women who are surgically candidate for myomectomy
* Age > 20 years

Exclusion Criteria:

* Contraindications for laparoscopic surgery and/or general anesthesia.
* Greater than five fibroids sized of 3cm or more
* Uterus extending beyond the umbilicus
* Major medical comorbidity or psychiatric illness, which could affect follow-up and/or compliance
* Patients undergoing concomitant complex surgical procedures at the time of myomectomy (such as resection of severe endometriosis etc.)
* Pregnancy
* Patients with any suggestion of malignancy in the pelvis
* Patients with cooperation of another main surgical procedures such as severe adhesiolysis or low anterior resection
* Patients who are severely anemic or who have significant medical conditions such as cardiac or pulmonary disease
* Patients who refuse to participate or give consent to the procedures

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myoma which are surgically candidate at educational hospitals
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Technical feasibilities and postoperative morbidity after E-NOTES for Myomectomy with Traction of Multidirectional Sutures | Postoperative surveillance including pain evaluation as routine clinical practise for 1 months
  Technical feasibility and postoperative morbidity will be evaluated in terms of overall or institutional conversion rate to convetional multi-port laparoscopy or laparotomy, operation time for each surgical procedures: dissection, morecellation, suturing, and total surgical procedures, complication, change of hemoglobin, and estimated blood loss

SECONDARY OUTCOMES:
Postoperative pain after E-NOTES for Myomectomy with Traction of Multidirectional Sutures by clinical variables such as incision size, type of port, size and number of myoma, or operation time. | Preoperative and postoperative pain
  Visual analogue scale will be used for pain evaluation: preoperative, postoperative 24 hour, postoperative 48 hour, postoperative 10 day (7 to 10 day), and postoperative 28 day (21 to 35 day).

CONTACTS AND LOCATIONS:
Overall Officials: Myong Cheol Lim, MD, PhD, Principal Investigator — National Cancer Center
Locations (2):
- South Korea (2):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - National Cancer Center, Koyang-si